CLINICAL TRIAL: NCT03562013
Title: Family Experience of Home Opioid Use After Pediatric Surgery: a Pilot Study
Brief Title: Family Experience of Home Opioid Use After Pediatric Surgery
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Conor McDonnell, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000060801
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A systematic review examining outpatient opioid use identified only three pediatric studies published between 2015 and 2016. Of these three, two studies had a short-term follow up with patients at three days after discharge; moreover, these three studies were limited by focusing on one surgical population, restriction of data to 0-12 yr old participants, and the other being a brief report. As a result, there are no pediatric studies that have examined opioid use amongst 0-18 yr olds, across multiple surgery types, and beyond 3 days after discharge.

DETAILED DESCRIPTION:
This study is being done to learn how long children (0-18 yrs) needed to use the prescribed opioid medication for and how families can be better prepared to provide adequate and safe pain management at home. Follow up will take place 28 days after discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Families are filling a prescription for opioid medications at Shoppers Drug Mart at The Hospital for Sick Children
* Parent has strong command of the English language (i.e., no interpreter required)

Exclusion Criteria:

* Child has used opioid medication at home within 6 months before the date of their surgical procedure
* Child has history of chronic pain
* Child is being discharged to a rehabilitation facility anticipated

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Any child (0-18 years) who has undergone a surgical procedure at The Hospital for Sick Children within 7 days of discharge.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire on Opioid use | 28 days following discharge from hospital
  Questionnaire on how families provide adequate and safe pain management at home

CONTACTS AND LOCATIONS:
Overall Officials: Conor Mc Donnell, MD, Principal Investigator — Staff Anesthesiologist
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Feinberg AE, Chesney TR, Srikandarajah S, Acuna SA, McLeod RS; Best Practice in Surgery Group. Opioid Use After Discharge in Postoperative Patients: A Systematic Review. Ann Surg. 2018 Jun;267(6):1056-1062. doi: 10.1097/SLA.0000000000002591. PMID 29215370
- [Derived] Caldeira-Kulbakas M, Stratton C, Roy R, Bordman W, Mc Donnell C. A prospective observational study of pediatric opioid prescribing at postoperative discharge: how much is actually used? Can J Anaesth. 2020 Jul;67(7):866-876. doi: 10.1007/s12630-020-01616-5. Epub 2020 Mar 12. PMID 32166621